CLINICAL TRIAL: NCT06641128
Title: Clinical Study Evaluating the Possible Efficacy and Protective Effect of Empagliflozin in Rheumatoid Arthritis Patients Treated with Methotrexate
Brief Title: The Possible Efficacy and Protective Effect of Empagliflozin in Rheumatoid Arthritis Patients Treated with Methotrexate
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nehad Waleed Karam, Pharmacist and Master's degree student, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Effect of Empagliflozin in RA
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA); Methotrexate Induced Nephrotoxicity; Methotrexate Adverse Reaction
Keywords: Rheumatoid Arthritis; Methotrexate side effect; empagliflozin role in RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MTX SC or IM - Empa tab (Active Comparator): IM or SC Methotrexate plus Empa tablets 25 mg once dailyf or 3 months.
  Interventions: Drug: MTX SC or IM; Drug: Empagliflozin 25mg tab
- MTX SC or IM - placebo tab (Placebo Comparator): IM or SC Methotrexate plus placebo tablet once daily for 3 months.
  Interventions: Drug: MTX SC or IM

INTERVENTIONS:
Drug: MTX SC or IM — IM or SC Methotrexate
Drug: Empagliflozin 25mg tab — Empa tablets 25 mg once daily for 3 months.
  Arms: MTX SC or IM - Empa tab

SUMMARY:
The primary aim of this clinical trial is to Evaluate the Possible Efficacy and Protective Effect of Empagliflozin in Rheumatoid Arthritis Patients Treated with Methotrexate.

Methodology:

This is a randomized, double blind placebo controlled parallel study that will be conducted on 44 patients with active rheumatoid arthritis.

Group1 (placebo group; n=22) which will receive IM or SC Methotrexate plus placebo tablet once daily for 3 months.

Group2 (Empa group; n=22) which will receive IM or SC Methotrexate plus Empa tablets 25 mg once daily for 3 months.

Duration: 3 months

Monitoring:

Participants will be followed up by weekly telephone calls and monthly direct meeting at scheduled visits to assess their adherence and to report any drug related adverse effects.

In summary, this clinical trial is designed to determine if empagliflozin is a safe and effective treatment for Rheumatoid Arthritis Patients Treated with Methotrexate by comparing its effects to a placebo and closely monitoring participants throughout the study.

DETAILED DESCRIPTION:
Increasing evidence suggests that the nucleotide-binding domain, leucine-rich-containing family, pyrin domain-containing-3 (NLRP3) inflammasome is involved in the pathogenesis of RA. Anti-citrullinated protein antibodies (ACPA) are a group of autoantibodies against citrullinated proteins/peptides and are biomarkers of RA. ACPA promotes IL-1 production in rheumatoid arthritis by activating the NLRP3 inflammasome. Several studies have shown an upregulation of NLRP3 mRNA and NLRP3-associated proteins in monocytes, macrophages, and dendritic cells in RA patients. Polymorphisms in the NLRP3 gene indirectly reflect the susceptibility, disease severity and treatment effect of RA .

Methotrexate (MTX) is a folic acid antagonist-an antiproliferative drug, as it is known. MTX is a gold-standard antirheumatic agent in the treatment of rheumatoid arthritis, Various side effects may occur during the treatment of inflammatory diseases, ranging from mild to severe side effects and even leading to treatment discontinuation .

The complications of chronic MTX toxicity include kidney injury, hepatotoxicity, mucositis, neurotoxicity, hyperglycemia, hematologic complications and myelosuppression . Chronically MTX-poisoned patient is the one with a long-standing RA or psoriasis/psoriatic arthritis presenting with sudden onset of erosions or ulcers in psoriatic plaques and/or sudden onset of severe mucosal ulceration in the oral cavity with or without diarrhea and fever secondary to infection. Mucosal ulceration was seen in most chronic cases.

The reason that MTX-induced renal dysfunction is a fundamental problem is that renal function in RA patients is already compromised. Because the renal tubules excrete more than 90% of MTX. MTX toxicity is enhanced by drugs that reduce renal elimination, including sulfonamides, aminoglycosides, cisplatin, penicillins, and colchicine, as well as by drugs that displace methotrexate from protein binding sites in plasma, including sulfonamides, phenytoin, retinoids, and barbiturates .

Gastrointestinal side effects of MTX is the main dose-limiting issue for the use of MTX is gastrointestinal toxicity.

MTX has been elucidated to exhibit a negative effect on the mitochondrial respiratory chain and hence induce excessive production of reactive oxygen species (ROS) leading to oxidative stress . ROS can initiate cellular macromolecule damage and induce lipid peroxidation leading to cell death . MTX showed a significant increase in liver lipid peroxidation indicator (Malondialdehyde) in rats. Therefore, attenuating the formation of ROS and inhibiting oxidative stress has been introduced as a suitable option to protect the organ against MTX-induced toxicity.

Empagliflozin (Empa) belongs to a novel class of anti-hyperglycemic drugs which was approved by the FDA on August 1, 2014. Contrary to conventional hypoglycemic agents, Empa lowers blood glucose by inhibiting the activity of sodium-glucose cotransporter-2 (SGLT-2) in proximal renal tubules. The SGLT2 transporter is mostly expressed in the proximal tubules in the kidney but is found also in other organs, such as the liver, thyroid, muscle, and heart. The receptor's function is to reabsorb glucose coupled with sodium ion from the excreted urine back to the blood .

Apart from glucose lowering, Empa has other pleiotropic effects and antioxidant effects. These benefits lead to cardiovascular protection through decreasing weight, lowering blood pressure, increasing the elasticity of the arteries, and reducing its stiffness, lowering lipid production, decreasing systemic inflammation and the release of inflammatory biomarkers, increasing insulin production, decreasing insulin resistance, and decreasing uric acid levels . Furthermore, different studies have elucidated that Empa exerts beneficial roles in the brain, peripheral neurons, kidneys, liver, and gastrointestinal tract .

Empa reduced proinflammatory cytokines such as interleukin-1β (IL-1β) , IL-6 and IL-8 in doxorubicin-treated mice model through affecting the expressions of NLRP3 and MyD88 related pathways which are also involved in pathophysiology of rheumatoid arthritis .

Several studies have shown the protective effects of Empa on different liver-related pathologies induced by ethanol and high-fat diets in rats. Regarding the possible molecular mechanisms of Empa, attenuation of oxidative stress has been presented as the underlying mechanism. It has been reported that the protective effects of Empa are associated with its ability to reduce ROS generation and induction of cellular antioxidant defense. In rats, Empa increase activity of superoxide dismutase (SOD), catalase (CAT) and glutathione peroxidase (GPX) which are a first line antioxidant defense system .

Several studies showed that marked increase in both alanine transaminase (ALT) and aspartate transaminase (AST) serum concentrations in patients treated with MTX. However, Empa treatment significantly reduced the elevation of serum concentrations of AST and ALT induced by MTX in rats .Aim of the study This study aimed to investigate the possible efficacy and protective effect of Empagliflozin in rheumatoid arthritis patients treated with methotrexate.

Patients and method

Study design and study population:

The patients will be recruited from Outpatient Clinic of Internal Medicine, Rheumatology and Immunology Department, Mansoura University Hospital, Mansoura, Egypt. The study duration will be 3 months. The blindness will be maintained by the similarity between the placebo and Empa tablets. The patients will be randomized using sealed envelope method with assigned code into two groups

Ethical approval:

The study will be conducted following the ethical standards of Helsinki declaration in 1964 and its later amendments. The study will be approved by the Research Ethics Committee of Tanta University and Mansoura University. The study will be registered as a clinical trial on ClinicalTrials.gov. All participants will be informed about the benefits and risks of the study. Any unexpected risks that will appear during the research will be clarified to the participant and to the concerned ethical committee on time. The privacy of all participants will be respected, and all data will be confidential. A written informed consent will be obtained from all patients (or their caregivers if the patient is unable to write or is cognitively impaired). The study will be conducted between 2024 - 2026.

Inclusion criteria:

Patients with active rheumatoid arthritis (not in remission) according to 28 joints disease activity score (DAS-28) >2.6 (Aletaha et al., 2010).

Age range between 18 and 60 years old. Both sexes. Body mass index (BMI), age, disease activity, and disease duration matched patients.

Patients receive methotrexate and other conventional DMARDs.

Exclusion criteria:

Patients with renal or hepatic diseases (chronic liver disease, liver cirrhosis, alcoholic hepatitis, or chronic alcoholism).

Patients receiving biological DMARDs during 4 weeks before the first dose of Empa.

Patients with hypersensitivity to study medications. Patients using antioxidants except Empa. Pregnant and lactating females. Pre-existing blood disorders, such as bone marrow hypoplasia, leukopenia, thrombocytopenia, or significant anemia.

Patient with HIV/AIDS, blood dyscrasias, or radiotherapy.

Methods:

All participants included in this study will be subjected to the following:

History, demography, and anthropometric data collection All participants will be submitted to physical and clinical examination, demographic data collection (age, sex, and history) and measurement of weight and height with subsequent calculation of body mass index according to the following formula: BMI=[weight (Kg)÷〖height〗^2 (m^2 )].

Blood sample collection and biological assessment Before and 3 months after the intervention, 10 ml of venous blood will be withdrawn by antecubital venipuncture from each participant after overnight fasting (10-12 h fasting period) between 8:30 and 10:30 am. 5 ml of blood will be used for evaluation of the following parameters.

Routine laboratory tests Erythrocyte sedimentation rate (ESR) C-reactive protein (CRP) Rheumatic factor (RF) Liver function test Kidney function test

Then the remaining 5 ml of blood will be transferred into a plain test tube and centrifuged at 3000 rpm for 10 min and then serum samples will be kept frozen at -80 C until analysis of biological markers:

NOD-like receptor protein 3 (NLRP3) Interleukin-1β (IL-1β) Superoxide dismutase (SOD) Clinical assessment Before and 3 months after the intervention, calculation of 28-joint count Disease Activity Score (DAS28) using C-reactive protein (CRP (where high disease activity ≥ 5.1, low disease activity ≤ 3.2, and remission <2.6.

Assessment of participants' adherence, side effects and tolerability Empa and placebo tablets will be provided on monthly intervals and the participants adherence will be assessed through counting the returned pills and through the medication refilling rate. Participants will be followed up by weekly telephone calls and monthly direct meeting at scheduled visits to assess their adherence and to report any drug related adverse effects. The adverse effects will be collected using adverse effect check list. Participant was considered non-adherent and excluded from the study if consumed less than 90% of the study medications or lost the follow-up meetings at any month of intervention.

Sample size calculation:

Using SPSS program version 25 (SPSS Inc, Chicago, IL, USA, 2017) and with the assumption of significance level of 0.05 (confidence interval of 95%) and statistical power of 80% which in turn will provide a large effect size of 0.80 to detect the difference in the outcome measured between the two groups using independent (Unpaired) t-test, the total sample size will be 36 patients in both arms (18 per group). Assuming that, the attrition rate is 20%, the total sample size will be 44 patients (22 patients per group).

Statistical analysis The collected data will be tabulated using Microsoft Office Excel, 2019 (Microsoft Corporation).

The statistical analysis will be performed using IBM SPSS Statistics version 28 software (IBM Corp, Armonk, NY, USA).

All graphs will be created with graph Pad prism 6.01 software (Graph pad Software, La Jolla CA, USA).

Data will be tested for normality using Shapiro-Wilk test or Kolmogorov-Smirnov test.

Parametric data will be analyzed using Paired and Un-Paired t-test to compare the means within the same group and to compare the means of the two groups respectively.

Non- Parametric data will be analyzed using Mann Whitney U test to compare the means within the same group and to compare the means between groups.

Categorical data will be analyzed using Chi-Square test. Fisher's exact test will be used to analyses the reported adverse effects. Correlation between variables will be assessed using Pearson or Spearman correlation coefficient which appropriate.

Data will be expressed as the mean ± SD, medians, range, number, and percent as appropriate.

The significance level will be set at p≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with active rheumatoid arthritis (not in remission) according to 28 joints disease activity score (DAS-28)
* Age range between 18 and 60 years old.
* Both sexes.
* Body mass index (BMI), age, disease activity, and disease duration matched patients.

Exclusion Criteria:

* Patients with renal or hepatic diseases (chronic liver disease, liver cirrhosis, alcoholic hepatitis, or chronic alcoholism).
* Patients receiving biological DMARDs during 4 weeks before the first dose of Empa.
* Patients with hypersensitivity to study medications.
* Patients using antioxidants except Empa.
* Pregnant and lactating females.
* Pre-existing blood disorders, such as bone marrow hypoplasia, leukopenia, thrombocytopenia, or significant anemia.
* Patient with HIV/AIDS, blood dyscrasias, or radiotherapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
calculation of DAS28-CRP score for measure disease activity | From enrollment to the end of treatment at 3 months
  this is a score for measure of disease activity in RA ; 2.6 mean RA is in remission 2.6 to 3.2 mean low level of disease activity More than 3.2 mean active disease that may require change in medication More than 5.1 mean very active disease that requires careful monitoring and adjustment to medication

SECONDARY OUTCOMES:
measurement of the levels of Interleukin-1β and Superoxide dismutase | From enrollment to the end of treatment at 3 months
  The inflammatory cytokine interleukin 1 (IL 1) is a key mediator in the autoimmune disease rheumatoid arthritis (RA) Superoxide dismutase as antioxidant regulates oxidative stress and lipid metabolism

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Internal Medicine, Rheumatology and Immunology Department, Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McInnes IB, Schett G. The pathogenesis of rheumatoid arthritis. N Engl J Med. 2011 Dec 8;365(23):2205-19. doi: 10.1056/NEJMra1004965. No abstract available. PMID 22150039
- [Background] Yin H, Liu N, Sigdel KR, Duan L. Role of NLRP3 Inflammasome in Rheumatoid Arthritis. Front Immunol. 2022 Jun 27;13:931690. doi: 10.3389/fimmu.2022.931690. eCollection 2022. PMID 35833125
- [Background] Kalantari E, Zolbanin NM, Ghasemnejad-Berenji M. Protective effects of empagliflozin on methotrexate induced hepatotoxicity in rats. Biomed Pharmacother. 2024 Jan;170:115953. doi: 10.1016/j.biopha.2023.115953. Epub 2023 Dec 7. PMID 38064971
- [Background] Guo Q, Wang Y, Xu D, Nossent J, Pavlos NJ, Xu J. Rheumatoid arthritis: pathological mechanisms and modern pharmacologic therapies. Bone Res. 2018 Apr 27;6:15. doi: 10.1038/s41413-018-0016-9. eCollection 2018. PMID 29736302
- [Background] Quagliariello V, De Laurentiis M, Rea D, Barbieri A, Monti MG, Carbone A, Paccone A, Altucci L, Conte M, Canale ML, Botti G, Maurea N. The SGLT-2 inhibitor empagliflozin improves myocardial strain, reduces cardiac fibrosis and pro-inflammatory cytokines in non-diabetic mice treated with doxorubicin. Cardiovasc Diabetol. 2021 Jul 23;20(1):150. doi: 10.1186/s12933-021-01346-y. PMID 34301253
- [Background] Theofilis P, Sagris M, Oikonomou E, Antonopoulos AS, Siasos G, Tsioufis K, Tousoulis D. Pleiotropic effects of SGLT2 inhibitors and heart failure outcomes. Diabetes Res Clin Pract. 2022 Jun;188:109927. doi: 10.1016/j.diabres.2022.109927. Epub 2022 May 14. PMID 35577035
- [Background] Gagnon KB, Delpire E. Sodium Transporters in Human Health and Disease. Front Physiol. 2021 Feb 25;11:588664. doi: 10.3389/fphys.2020.588664. eCollection 2020. PMID 33716756
- [Background] Kolli VK, Natarajan K, Isaac B, Selvakumar D, Abraham P. Mitochondrial dysfunction and respiratory chain defects in a rodent model of methotrexate-induced enteritis. Hum Exp Toxicol. 2014 Oct;33(10):1051-65. doi: 10.1177/0960327113515503. Epub 2013 Dec 17. PMID 24347301